CLINICAL TRIAL: NCT00713401
Title: An Open-Label, Sequential-Group, Dose-Escalation Study To Evaluate The Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous Tecadenoson Alone and in Combination With a Beta-Blocker in Adults With Rapid Atrial Fibrillation (CVT 4129)
Brief Title: Safety Study of Tecadenoson to Treat Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVT 4129
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — tecadenoson; esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort A (Experimental): Period 1: 75 mcg, i.v. bolus. Period 2: 75 mcg, i.v. bolus + esmolol low dose infusion
  Interventions: Drug: Tecadenoson; Drug: Esmolol
- Cohort B (Experimental): Period 1: 150 mcg, i.v. bolus. Period 2: 150 mcg, i.v. bolus + esmolol low dose infusion
  Interventions: Drug: Tecadenoson; Drug: Esmolol
- Cohort C (Experimental): Period 1: 300 mcg, i.v. bolus. Period 2: 300 mcg, i.v. bolus + esmolol low dose infusion
  Interventions: Drug: Tecadenoson; Drug: Esmolol
- Cohort D (Experimental): Period 1: 75 mcg, i.v. bolus. Period 2: 75 mcg, i.v. bolus + esmolol high dose infusion
  Interventions: Drug: Tecadenoson; Drug: Esmolol
- Cohort E (Experimental): Period 1: 150 or 300 mcg, i.v. bolus. Period 2: 150 or 300 mcg, i.v. bolus + esmolol high dose infusion
  Interventions: Drug: Tecadenoson; Drug: Esmolol

INTERVENTIONS:
Drug: Tecadenoson — Tecadenoson administered intravenously (i.v.)
  Other Names: CVT-510
Drug: Esmolol — Esmolol low dose infusion according to manufacturer's instructions
  Other Names: Brevibloc®

SUMMARY:
Assess the tolerability and safety of a rapid bolus of tecadenoson at different dose levels when given alone and in combination with a beta-blocker (esmolol) in patients with atrial fibrillation to control rapid heart rate. Explore the pharmacokinetic and pharmacodynamic effects when given alone and in combination with beta-blocker (esmolol).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of atrial fibrillation in need of treatment for rate control
* Be able and willing to abstain from any antiarrhythmics, including atrioventricular (AV) nodal blocking agents (except for esmolol per protocol), from no later than 8:00 p.m. on the day prior to dosing until completion of the last dose period assessment
* Be able and willing to abstain from xanthine- or chocolate-containing foods, beverages, and medications
* Females must be post-menopausal or sterilized; or if of childbearing potential, must not be breastfeeding and must have a negative pregnancy test at screening and no intention of becoming pregnant during the course of the study. Males and females must be using adequate contraception during the study.

Exclusion Criteria:

* Have a known accessory pathway
* Have active myocardial ischemia or recent acute coronary syndrome
* Have acute or overt heart failure, bradycardia, heart block greater than first degree, or cardiogenic shock
* Have allergies or contraindications to treatment with esmolol or aminophylline, or any of their constituents
* Have a supine cuff systolic blood pressure < 90 mm Hg
* Be undergoing treatment with theophylline/aminophylline preparations, Trental® (pentoxifylline), or carbamazepine
* Have asthma or other reactive airways disease currently on-treatment
* Have a history of an active or chronic pancreatic disease or clinically significant increased levels of serum amylase or lipase

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced Adverse Events (AEs) and Graded Laboratory Abnormalities | Baseline to Day 7

SECONDARY OUTCOMES:
Change in cardiac parameters R-R interval and ventricular rate measured by electrocardiogram | Baseline to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- CV Therapeutics, Inc., Palo Alto, California, United States

REFERENCES:
- [Derived] Corino VD, Holmqvist F, Mainardi LT, Platonov PG. Beta-blockade and A1-adenosine receptor agonist effects on atrial fibrillatory rate and atrioventricular conduction in patients with atrial fibrillation. Europace. 2014 Apr;16(4):587-94. doi: 10.1093/europace/eut251. Epub 2013 Aug 29. PMID 23989533